CLINICAL TRIAL: NCT00235118
Title: An Evaluation of the Safety and Effectiveness of the Cordis Bilateral AAA Device Compared to Open Surgical Repair for the Treatment of Abdominal Aortic Aneurysm
Brief Title: Cordis Bilateral AAA Device Compared to Open Surgical Repair of Abdominal Aortic Aneurysms (ARIBA)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P98-4601
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2005-12-09 (Estimated); Status verified 2005-10

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

INTERVENTIONS:
Device: Cordis AAA Bilateral Device

SUMMARY:
The objective of this study is to assess the safety and effectiveness of the Cordis Bilateral AAA device and its Delivery System compared to open surgical repair for the treatment of Abdominal Aortic Aneurysm (AAA).

ELIGIBILITY:
Inclusion Criteria:

- Anatomic (stent-graft)

Aortic Aneurysm Diameter

* > 4.5 cm
* Those aortic aneurysms < 4.5 cm that are at least 1.5 times the diameter of the aorta with a size increase of 5 mm or greater over a six month period will also be included for possible treatment.
* Aorto-iliac aneurysms in which the aortic aneurysm is < 4.5 cm but the iliac artery aneurysms are > 3.0 cm in diameter or there is evidence of recent expansion (5 mm or greater over a six month period) in iliac aneurysms < 3.0 cm.
* Saccular aortic aneurysms > 3.0 cm.

Aortic Neck

* Diameter > 17 mm and < 28 mm (Phase I)
* Diameter > 14 mm and < 28 mm (Phase II)

Angulation Neck Length < 45° > 15 mm <60° > 25 mm

Iliac Arteries

* Diameter > 8 mm and < 18 mm (Phase I and Phase II)
* At least one common iliac artery with a cuff > 15 mm.

Diameter Aortic Neck Common Iliac 26-28 mm 13-18 mm 23-25.9 mm 10-17 mm 20-22.9 mm 9-15 mm 17-19.9 mm 8-13 mm 14-16.9 mm 8-11mm

*NOTE: An aortic diameter cannot be treated if the iliac diameter is not in the same range (e.g. 26-28 mm aortic necks must be in conjunction with 13-18 mm common iliacs).

Anatomic (surgical controls)

· Surgical controls will be required to meet only the aortic or aorto-iliac aneurysm size requirements for anatomic inclusion criteria.

Aortic Aneurysm Diameter

* > 4.5 cm
* Those aortic aneurysms <4.5 cm that are at least 1.5 times the diameter of the aorta with a size increase of 5 mm or greater over a six month period will also be included for possible treatment.
* Aorto-iliac aneurysm in which the aortic aneurysm is <4.5 cm but the iliac artery aneurysm are >3.0 cm in diameter or there is evidence of recent expansion (5 mm or greater over a six month period) in iliac aneurysms <3.0 cm.
* Saccular aortic aneurysms > 3.0 cm.
* Clinical (stent-graft)
* Males and non-pregnant females > 40 years of age.
* Clinical (surgical controls)

Surgical control patients will be required to meet all of the above-stated stent-graft clinical inclusion criteria.

Exclusion Criteria:

Anatomic (stent-graft)

Aortic Aneurysm Diameter

· < 4.5 cm that are not at least 1.5 times the diameter of the aorta with evidence of a size increase of 5 mm or greater within a six month period.

Aorto-iliac Aneurysms

* < 3.0 cm in diameter unless evidence of recent expansion (5 mm or greater within a six month period).
* The iliac portion of the aneurysm extending to the bifurcation bilaterally which would necessitate covering both internal iliac arteries with the device.

Aortic Neck

* Diameter < 17 mm and > 28 mm (Phase I)
* Diameter < 14 and >28 (Phase II)
* Thrombus lined
* Highly calcified

  * NOTE: See inclusion criteria for length below the renals and degree of angulation.

Iliac Arteries

* < 8 mm and > 18 mm (native) (Phase I and Phase II)
* Highly calcified (common)
* Neither common iliac artery with a cuff > 15 mm.

  * NOTE: See inclusion criteria for aortic neck and iliac artery diameters.

Anatomic (surgical controls)

· Surgical controls will be excluded based only on the aortic or aorto-iliac aneurysm size requirements for anatomic exclusion criteria.

Aortic Aneurysm Diameter

· < 4.5 cm that are not at least 1.5 times the diameter of the aorta with evidence of a size increase of 5 mm or greater within a six month period.

Aorto-Iliac Aneurysms

* < 3.0 cm in diameter unless evidence of recent expansion (5 mm or greater within a six month period).
* The iliac portion of the aneurysm extending to the bifurcation bilaterally which would necessitate surgically covering both internal iliac arteries.

Clinical (stent-graft)

1. Ruptured abdominal aortic aneurysm.
2. Renal insufficiency - creatinine level > 2.5 mg/dl.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29
Dates: Start 1999-12; Study Completion 2006-02

PRIMARY OUTCOMES:
Primary success is defined as freedom from all of the following: rupture of aneurysm, enlargement of aneurysm > 0.5 cm on CT scan, with or without endoleak, as compared to any previous measurement, symptomatic aneurysm requiring treatment.
The absence of major complications at thirty days defined as arterial thrombosis, respiratory impairment, renal failure, myocardial infarction (M.I.) and stroke in combination with the absence of major complications at one year.

SECONDARY OUTCOMES:
· Technical success defined as the successful access and deployment of the device at the appropriate anatomic location with aneurysmal exclusion determined by angiography at the time of deployment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Marin, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mt. Sinai Hospital, New York, New York, United States